CLINICAL TRIAL: NCT02903043
Title: Expression of miR-204 and Consequences on Capillarization in Limb Muscles of Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Expression of miR-204 and Consequences on Capillarization in Limb Muscles of Patients With COPD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Annie Dubé, Ph.D., Laval University
Other Study IDs: MIR-20895
Record Dates: First submitted 2015-04-09; First posted 2016-09-16 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: MicroRNAs; Angiogenesis; Skeletal muscle; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Blood sample ad muscle biopsy of vastus lateralis (quadriceps)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- COPD patients: Quadriceps biopsies will be done. No drug administration.
- Healthy controls: Quadriceps biopsies will be done. No drug administration.

SUMMARY:
Limb muscle dysfunction, characterized by loss of capillaries, is amongst the most troublesome systemic consequences of chronic obstructive pulmonary disease (COPD) leading to poor functional status and premature mortality.

One prevailing hypothesis stipulates that modification in the expression of miR-204 leads to change the regulation of angiogenesis in vastus lateralis of patients with COPD when compared to controls.

DETAILED DESCRIPTION:
The investigators objective is to investigate the impact of COPD on key signaling pathways involved in the muscle angiogenesis. Mild to severe COPD patients and healthy controls will be recruited. All of the investigators patients will undergo a thorough baseline assessment in pulmonary capacity and body composition. Blood sampling and biopsy of the quadriceps will be done. Key proteins and microRNAs of signaling intramuscular pathways involved in angiogenesis will be measured in the quadriceps.

ELIGIBILITY:
Inclusion Criteria:

* COPD (FEV1/FVC < 0.70)
* Healthy subjects: no evidence of airways obstruction (FEV1/FVC > 0.70 and FEV1 > 0.80 predicted)
* Smoking history > 10 pack-years
* Ex-smoker >6 months

Exclusion Criteria:

* Chronic hypoxemia and/or hypercapnia (PaO2 < 60 mmHg or SpO2 < 88% at rest and/or PaCO2 > 45 mmHg)
* Recent exacerbation or oral corticosteroids (< 2 months)
* Recent cancer (< 3 years)
* Diabetes
* Myopathy, neuromuscular, neurological or articular diseases
* Kidney disease
* Other respiratory diseases
* Unstable cardiac disease
* Physical activity score > 9 in the Voorips questionnaire
* BMI > 30

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with COPD
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-04 (Actual); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
miR-204 in limb muscles in patients with COPD | At baseline (COPD patients in a stable state of the disease)
  i)To measure miR-204 level in the quadriceps of patients with COPD in comparison to controls.
  ii) To study possible involvement of miR-204 on pathways regulating angiogenesis and on muscle microcirculation in these individuals.

SECONDARY OUTCOMES:
microRNAs in limb muscles of patients with COPD | At baseline (COPD patients in a stable state of the disease)
  i) To measure microRNAs levels in the quadriceps of patients with COPD in comparison to controls.
  ii) To study possible involvement of these microRNAs on pathways regulating myogenesis, angiogenesis and on muscle microcirculation in these individuals.

CONTACTS AND LOCATIONS:
Overall Officials: François Maltais, MD, Study Director — Laval University
Locations (1):
- Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Canada

IPD SHARING:
Plan to Share IPD: Undecided